CLINICAL TRIAL: NCT04247217
Title: Prostate Cancer Immune Profiling Before, During and After HDR-brachytherapy in Local Relapsed Prostate Cancer (PRIMUS-study)
Brief Title: Immune Profiling After HDR in Local Relapsed Prostate Cancer
Acronym: PRIMUS
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: PRIMUS
Record Dates: First submitted 2020-01-17; First posted 2020-01-29 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer; PD-L1
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In patients receiving HDR salvage brachytherapy for locally relapsed prostate cancer serial biopsies will be performed at 4 different time points. Furthermore, peripheral blood samples during anesthesia will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: HDR salvage brachytherapy — In patients receiving HDR salvage brachytherapy for locally relapsed prostate cancer serial biopsies will be performed at 4 different time points.
  Other Names: biopsies

SUMMARY:
Immunotherapy is currently revolutionizing the field in oncology. However, prostate cancer until now fails to respond to classical IO, like PD-1 and CTLA-4 inhibitors. Radiotherapy (RT) delivered to the primary tumor impacts both tumor cells and surrounding stromal cells. Radiation damage to cancer cells exposes tumor-specific antigens leading to increased visibility to the immune system by improved priming and activation of cytotoxic T cells. RT-induced modulation of the tumor microenvironment may also facilitate the recruitment and infiltration of immune cells by increasing the expression or T-cell attracting chemokines and by increasing T-cell docking molecules on the endothelial cells like VCAM-1. The main-hypothesis is that HDR-brachytherapy will turn an immunologically "cold" (no T-cell infiltrations) prostate cancer into an immunologically "hot" (CD4 and CD8-cell infiltrations) tumor, creating leverage points for different forms of IO.

DETAILED DESCRIPTION:
Prospective analysis of biopsies from 10 patients with local recurrence in the prostate selected for salvage HDR brachytherapy in MAASTRO Clinic, Maastricht. HDR treatment is standard in Maastro Clinic for local relapses of prostate cancer after previously irradiation (internal or external).

Biopsies will be taken at 4 different time points (before and after the 1st fraction; before the 2nd and 3rd fraction of the salvage treatment).

Several immunotyping (expression of PD-(L)-1, CXCL12, IL-23 receptor, etc.) and HLA class I expression will be performed on the biopsies. In addition, HLA genotypes will be determined on DNA isolated from pheripheral blood.

The plasma and the biopsies will be stored for eventually additional research.

ELIGIBILITY:
Inclusion Criteria:

* Local relapse of prostate cancer, who is candidate for a salvage HDR treatment:
* Biochemical relapse (PSA increase)
* Local relapse on imaging: PSMA scan, mp-MRI
* Pathology proven relapse

  * Willing and able to comply with the study prescriptions.
  * 18 years or older
  * Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Not eligible for proposed (HDR brachytherapy) treatment:

  * Life expectancy < 10 years
  * Distant Metastasis
  * Recently TURP with big urethral defect
  * Not able to stop anticoagulants
  * Flow < 10 ml/sec • No compliance to study procedure

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate tumor biopsies
Study Population: Patients with local relapse of prostate cancer, who are candidate for a salvage HDR treatment will be asked to participate in this study at the time of intake.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Expression of PD-(L)-1 receptor | up to 28 days
  Expression of PD-(L)-1 receptor induced by HDR-brachytherapy in prostate tumor biopsies of local relapses of prostate cancer of 10 patients at 4 different time points.

SECONDARY OUTCOMES:
Expression patterns of CXCL12 | up to 28 days
  Expression of CXCL12 receptor induced by HDR-brachytherapy in prostate tumor biopsies of local relapses of prostate cancer of 10 patients at 4 different time points
Expression patterns of IL-23 | up to 28 days
  Expression of IL-23 receptor induced by HDR-brachytherapy in prostate tumor biopsies of local relapses of prostate cancer of 10 patients at 4 different time points
Expression patterns of MDSC | up to 28 days
  Expression of MDSC receptor induced by HDR-brachytherapy in prostate tumor biopsies of local relapses of prostate cancer of 10 patients at 4 different time points
Changes in T cell infiltration profiles | up to 28 days
  Changes in T cell infiltration profiles induced by HDR-brachytherapy in prostate tumor biopsies of local relapses of prostate cancer of 10 patients at 4 different time points
Changes in HLA class I-A expression on tumor cells | up to 28 days
  Changes in HLA class I-A expression on tumor cells induced by HDR-brachytherapy in prostate tumor biopsies of local relapses of prostate cancer of 10 patients at 4 different time points
Changes in HLA class I-B expression on tumor cells | up to 28 days
  Changes in HLA class I-B expression on tumor cells induced by HDR-brachytherapy in prostate tumor biopsies of local relapses of prostate cancer of 10 patients at 4 different time points
Changes in HLA class I-C expression on tumor cells | up to 28 days
  Changes in HLA class I-C expression on tumor cells induced by HDR-brachytherapy in prostate tumor biopsies of local relapses of prostate cancer of 10 patients at 4 different time points

CONTACTS AND LOCATIONS:
Overall Officials: Ben Vanneste, MD, PhD, Principal Investigator — Maastro
Locations (1):
- Maastro, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No